CLINICAL TRIAL: NCT05799378
Title: A Phase III, Randomized, Double-Blind Placebo-Controlled, Non-Inferiority, Multi-Center Study of the Effects of Stopping Hydroxychloroquine in Elderly Lupus Disease
Brief Title: Effects of Stopping Hydroxychloroquine in Elderly Lupus Disease
Acronym: SHIELD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-00071
Record Dates: First submitted 2023-03-23; First posted 2023-04-05 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Hydroxychloroquine; systemic lupus erythematosus; elderly lupus disease; lupus; sle; plaquenil
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Hydroxychloroquine (HCQ) (Experimental): Patients will receive a 90-day supply of HCQ at their screening visit, at 2 months, 4 months, 6 months, 8 months, and 10 months. All patients will return their current supply along with a completed dosing diary at each visit and receive a new supply in exchange. The HCQ dose administered will match each patient's dosage of HCQ at enrollment.
  Interventions: Drug: Hydroxychloroquine
- HCQ-Matching Placebo (Placebo Comparator): Patients will receive a 90-day supply of HCQ-matching placebo at their screening visit, at 2 months, 4 months, 6 months, 8 months, and 10 months. All patients will return their current supply along with a completed dosing diary at each visit and receive a new supply in exchange. The HCQ-matching placebo dose administered will match each patient's dosage of HCQ at enrollment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine 200mg capsules. Administered orally.
  Arms: Hydroxychloroquine (HCQ)
Drug: Placebo — Hydroxychloroquine-matching placebo capsule. Administered orally.
  Arms: HCQ-Matching Placebo

SUMMARY:
Hydroxychloroquine (HCQ) is a systemic lupus erythematosus (SLE) medication that has been very effective in reducing lupus disease activity and keeping patients stable with reduced symptoms. Despite a track record of safety with regard to infection compared to traditional immunosuppressive agents, the risk of HCQ retinal toxicity escalates with continued use. Evaluation using sensitive standard of care approaches suggests nearly a third of patients accrue retinal damage. Data are needed to accurately weigh the balance between accumulating ocular exposure of HCQ versus the risk of disease flare in a population that may have more inactive disease than younger patients. The purpose of this trial is to address the safety of withdrawal of HCQ in SLE patients =60 years old. The central hypothesis is that HCQ can be safely discontinued in stable/quiescent patients assessed by validated disease activity and flare instruments in the context of serologic, cytokine and transcriptomic profiling. Patients will be randomized to either the placebo or active arm and followed every 2 months for one year to assess disease activity and flares.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Age ≥ 60 years at time of enrollment
* Normal OCT and VF assessment within 6 months of screening visit
* Ability to take oral medication
* Have established SLE (≥ 4 ACR criteria or SLICC criteria or ≥ 10 points by EULAR criteria, SLE diagnosed at least seven years ago)
* Stable disease at screening visit by attaining DORIS remission (meeting all criterion listed below) and not on any immunosuppressants.

  * Criterion 1: Clinical SLEDAI= 0
  * Criterion 2: SELENA-SLEDAI PGA ≤ 0.5 (on a scale from 0-3, where 0 is no disease activity and 3 is maximum disease activity)
  * Criterion 3: Current prednisolone (or equivalent corticosteroid) dose ≤ 5 mg daily
* No moderate or severe flares one year prior to screening
* Taking ≥ 200 HCQ daily for ≥ 7 years

Exclusion Criteria:

* Any patient that does not attain stable disease status by DORIS
* Ophthalmologic evidence of retinopathy (these patients would be advised to discontinue HCQ and therefore unethical to randomize for this study)
* Clinical SLEDAI > 0
* Taking > 5 mg/day prednisone
* Taking any immunosuppressive drugs or biological agents (including: methotrexate, azathioprine, mycophenolate mofetil, mycophenolic acid, leflunomide, cyclosporine, cyclophosphamide, tacrolimus, rituximab, and belimumab)
* Any reason the treating rheumatologist is concerned about ongoing activity not captured by SLEDAI
* HCQ level < 100 ng/ml as this would support noncompliance and less reliance on HCQ to control activity
* Patient unwilling or unable to comply with study procedures for any reason
* Any indications of potentially diminished capacity, such as a diagnosis of dementia or cognitive impairment (including, but not limited to stroke-related cognitive impairment)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who Develop Moderate or Severe Flare based on the Revised SELENA SLEDAI Flare Index (rSFI) | Up to Month 12
  Number of participants who experience moderate or severe flares as defined by the rSFI.

SECONDARY OUTCOMES:
Number of Participants who Develop Moderate Flare based on rSFI | Up to Month 12
  Number of participants who experience moderate flares as defined by the rSFI.
Physician Global Assessment (PGA) Score at Month 12 | Month 12
  The Physician Global Assessment (PGA) of treatment response measures the overall response to treatment as assessed by the physician. The score ranges from +4 to (-4), where 4 = Markedly Improved, 0 = No change, and (-4) = markedly worse.
Number of Participants who Begin Prednisone Treatment | Up to Month 12
Number of Participants who Increase Prednisone Use | Up to Month 12
Number of Participants who Experience Thromboembolic Event | Up to Month 12
  Thromboembolic event includes, but is not limited to, venous thrombosis.
Number of Participants who Experience Cardiovascular Event | Up to Month 12
Number of Participants with New-Onset Diabetes | Up to Month 12
Number of Participants with New Retinal Toxicity | Up to Month 12
Change in 36-Item Short Form Survey Instrument (SF-36) Score | Baseline, Month 12
  The SF-36 is 36-item self-rated measure of quality of life. A scoring algorithm is used to convert the raw scores into a range from zero (the respondent has the worst possible health) to 100 where the respondent is in the best possible health.
Change in 29-Question Patient-Reported Outcomes Measurement Information System (PROMIS-29) Score | Baseline, Month 12
  PROMIS-29 consists of 29 questions rated on a scale from 1-5. The raw score is converted to a final T-score metric with a mean T-score of 50 and a standard deviation of 10. The final score ranges from 0 (worst possible outcome) to 100 (best possible outcome). The questionnaire assesses seven domains - depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, and ability to participate in social roles and activities.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Izmirly, Principal Investigator — NYU Langone Health; Jill Buyon, Principal Investigator — NYU Langone Health
Locations (10):
- United States (10):
  - University of California, Los Angeles, Los Angeles, California
  - Hackensack Meridian Health, Hackensack, New Jersey
  - VA NY Harbor Healthcare System, New York, New York
  - NYC Health + Hospitals/Bellevue, New York, New York
  - NYU Langone Health, New York, New York
  - Hospital for Special Surgery, New York, New York
  - Columbia University Irving Medical Center/New York Presbyterian, New York, New York
  - Montefiore Medical Center/Albert Einstein College of Medicine, The Bronx, New York
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Penn State MS Hershey Medical Center, Hershey, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared with investigators whose proposed use of the data has been approved by the co-PIs, Dr. Peter M. Izmirly and Dr. Jill P. Buyon, beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Peter.Izmirly@nyulangone.org and Jill.Buyon@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research. A copy of an informed consent form will also be made available.
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Investigators whose proposed use of the data has been approved by co-PIs, Dr. Peter M. Izmirly and Dr. Jill P. Buyon, will be granted access to the data to achieve aims outlined in the approved proposal. Requests should be directed to Peter.Izmirly@nyulangone.org and Jill.Buyon@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.